CLINICAL TRIAL: NCT06394063
Title: A Randomized, Double-blind, Placebo-controlled Trial of Efficacy and Safety of Low-dose Telitacicept for Prevention of Flares in SLE Patients With Low Disease Activity
Brief Title: Efficacy and Safety of Telitacicept for Prevention of Flares in SLE Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ttrial
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — telitacicept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telitacicept (Experimental): Telitacicept 160mg is administered subcutaneously every other week for 26 times on the background of standard therapy.
  Interventions: Biological: Telitacicept
- Placebo (Placebo Comparator): Placebo is administered subcutaneously every other week for 26 times on the background of standard therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Telitacicept — Telitacicept 160 mg SC every other week
  Arms: Telitacicept
Drug: Placebo — Placebo to Telitacicept
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled single-center clinical trial. The aim of this study is to investigate the efficacy and safety of low-dose telitacicept for prevention of flares in SLE patients with low disease activity.

DETAILED DESCRIPTION:
Background: There are still two major problems in the treatment of SLE: flare and long-term organ damage. BLISS-52 showed there was some reduction of flare (80% vs 71%) in belimumab , but the difference was not significant. Another study tested the efficacy and safety of atacicept for prevention of flares in patients with moderate-to-severe SLE in which analysis of atacicept 150 mg suggested benefit.

Telitacicept , a BAFF/APRIL dual-target-inhibitor, which has been proved to be effective in treatment of SLE. But there is no study to show its effectiveness for prevention of flares in SLE patients with low disease activity. In this study, we take telitacicept as maintain treatment in stable SLE patients to investigate the efficacy and safety of low-dose telitacicept for prevention of flares in SLE patients with low disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years;
2. SLE patients with low disease activity (SELENA-SLEDAI score< 8 at screening ); disease duration more than 3 months；no British Isles Lupus Assessment Group (BILAG) A and no more than one B;
3. A stable treatment regimen with fixed doses of prednisone (≤ 30mg/day), antimalarial, or immunosuppressive drugs (mycophenolate mofetil/azathioprine/ciclosporin /tacrolimus/methotrexate/leflunomide) for at least 3 months;
4. Sign the informed consent.

Exclusion Criteria:

1. Hepatic or renal dysfunction: alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) > 2 times upper normal limits; GFR < 60ml/min;
2. Exposure to cyclophosphamide within past 6 months before screening;
3. Exposure to any B cell targeted therapy (Rituximab/Belimumab/Telitacicept) within past 6 months before screening;
4. Pregnant women, lactating women;
5. History of Malignancy within the last 5 years, excluding adequately treated skin tumors (basal cell or squamous cell carcinoma) or carcinoma in situ of cervix;
6. Active hepatitis or a history of severe liver disease;
7. Current infections (HIV/tuberculosis/COVID-19, etc.) at screening;
8. A significant decrease in immunoglobulin level, IgG<5g/L;
9. Not suitable for the study in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with disease flares | 52 weeks
  Disease flare is defined by modified SELENA-SLEDAI SLE flare index (SFI).

SECONDARY OUTCOMES:
Percentage of patients with mild/moderate flares | 52 weeks
  Disease flare is defined by modified SELENA-SLEDAI SLE flare index (SFI).
Percentage of patients with major flares | 52 weeks
  Disease flare is defined by modified SELENA-SLEDAI SLE flare index (SFI).
Time to first disease flare | 52 weeks
  Time to first disease flare defined by modified SELENA-SLEDAI SLE flare index (SFI).
Prednisone dose at each visit | 52 weeks
  Compare the prednisone dose at each visit
PGA score at each visit | 52 weeks
  Compare the disease activity measured by PGA score at each visit
SELENA-SLEDAI score at each visit | 52 weeks
  Compare the disease activity measured by SELENA-SLEDAI score at each visit
Maintenance time of LLDAS/Remission | 52 weeks
  To record the maintenance time of LLDAS/Remission
Number of participants with adverse events as assessed by CTCAE v5.0 | 52 weeks
  The safety of telitacicept

OTHER OUTCOMES:
Subgroup analysis | 52 weeks
  Subgroup analysis aiming to investigate which population will benefit most from telitacicept with prespecified factors

CONTACTS AND LOCATIONS:
Locations (1):
- Ren Ji Hospital, Shanghai, China